CLINICAL TRIAL: NCT05576597
Title: A Pilot Study to Evaluate Efficacy and Safety of Butyrate Supplement in the Treatment of Rheumatoid Arthritis
Brief Title: Effect of Butyrate Supplement on Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ButyrateRA
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Butyric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Butyrate supplement (Experimental): 2 capsules butyrate supplement (containing 1200 mg of butyric acid ) once a day for 12 weeks Drug: sodium butyrate
  Interventions: Drug: Sodium Butyrate

INTERVENTIONS:
Drug: Sodium Butyrate — 2 capsules butyrate supplement once a day for 12 weeks

SUMMARY:
This study is a pilot study to evaluate the safety and efficacy of administering butyrate supplement on rheumatoid arthritis patients. Thirty participants will be included to receive butyrate supplement for 12 weeks. Changes of immune cell subtypes, markers of intestinal damage, intestinal flora and other laboratory indicators will be monitored.

DETAILED DESCRIPTION:
This is a single center, uncontrolled, open-label study to assess the efficacy and safety of butyrate supplement plus standard therapy in rheumatoid arthritis(RA). The patients will be given 2 sodium butyrate capsules (containing 1200 mg of sodium butyrate) daily as supplemental therapy. The objective is to assess the effects of 12 weeks of sodium butyrate supplementation on intestinal inflammation and immune regulation in patients with RA, specifically changes in T-cell subtypes and biomarkers associated with intestinal injury. Clinical manifestations and other laboratory indices will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age at the time of screening, weight≥35 kg.
* Diagnosed with rheumatoid arthritis satisfying the 1987 American College of Rheumatology classification criteria.
* Stable treatment, including DMARDs (disease-modifying anti-rheumatic drugs) and glucocorticoids, was stable in dose for at least 4 weeks, and no biological agents were used during the first 12 weeks of enrollment.
* Have given written informed consent

Exclusion Criteria:

* Patient presenting or having a history of other autoimmune diseases (such as Sjogren's syndrome, systemic lupus erythematosus, systemic sclerosis, vasculitis, etc.) and other arthritic diseases (such as spinal arthritis, psoriatic arthritis, reactive arthritis, etc.)
* Patient with ongoing or previous Stevens-Johnson syndrome, toxic epidermal necrolysis or erythema multiforme
* Patient with significantly impaired bone marrow function or significant anemia, leucopenia or thrombocytopenia induced by other disease
* Patient with persistent or severe infection within 3 months before enrollment
* Patient with uncontrolled hypertension, uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, terminal illness or other medical condition which would put the patient at risk of participating in the study according to the opinion of investigator
* Patient with cardiovascular, hepatic, neurological, endocrine, or other major systemic disease, which may make implementation of the protocol or interpretation of the study results difficult
* Patient who has severe hypoproteinemia (e.g., in case of severe liver disease or nephrotic syndrome), with serum albumin < 30 g/L)
* Patient who has moderate or severe impairment of renal function (the estimated glomerular filtration rate was < 60 mL/min/1.73 m2)
* Patient with impairment of liver function or persisting Alanine transaminase (ALT) or Aspartate aminotransferase (AST) elevations of more than 2-fold the upper limit of normal
* Patient with Known HIV positive status or positive serology for hepatitis B or C
* Pregnant or breastfeeding woman
* Women of childbearing potential
* Men wishing to father children during the course of the study or within the 24 months thereafter (or 3 months with the washout procedure)
* Patient with a congenital or acquired severe immuno-deficiency, a history of cancer or lymphoproliferative disease, or any patient who has received total lymphoid irradiation.
* Patient who enrolled in any other clinical trial involving off-label use of an investigational drug or device, or any other type of medical research
* Patient using any biologic agent such as anti-tumor necrosis factor, IL-6 receptor antagonist, anti-CD20 monoclonal antibody within 3 months prior to the first dose of treatment.
* Patient whose BMI (body mass index) is under 18.5 kg/m2 or more than 30 kg/m2
* Patient with history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Changes in disease Activity Score in 28 joints (DAS28) | Baseline,12 weeks
  Evaluating changes in DAS28 before and after treatment. DAS28 was calculated by the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (mm/h) or c-reactive protein (CRP) (mg/L), and patient's global assessment (PGA) of disease activity (based on the visual analog score [VAS], 0-100mm). Compared with the baseline, a lower DAS28 would mean an improvement in disease activity. Conversely, an increase in DAS28 indicates a deterioration in disease activity.

SECONDARY OUTCOMES:
Changes in the simplified disease activity index (SDAI) | Baseline and 12 weeks
  Evaluating changes in SDAI before and after treatment. The SDAI is a composite score based on the tender joints of 28 joints (TJC28), tender joints of 28 joints (SJC28), patients' and physicians' global assessments of disease activity (based on the visual analog score [VAS], 0-10cm), and c-reactive protein (CRP). Compared with the baseline, a lower SDAI would mean an improvement in disease activity. Conversely, an increase in SDAI indicates a deterioration in disease activity.
Changes in the clinical disease activity index (CDAI) | Baseline and 12 weeks
  Evaluating changes in CDAI before and after treatment. The Clinical Disease Activity Index (CDAI) is a composite score based on the TJC28, SJC28, and patients'and physicians'assessments (based on the visual analog score [VAS], 0-10cm). Compared with the baseline, a lower CDAI would mean an improvement in disease activity. Conversely, an increase in CDAI indicates a deterioration in disease activity.
Changes in T cell subtypes. | Baseline, 4 weeks and 12 weeks
  Evaluating changes in the percentage of T cell subtypes, especially T regulatory cells, in peripheral blood before and after treatment.
Changes in c-reactive protein (CRP). | Baseline, 4 weeks and 12 weeks
  Evaluating changes in concentration of CRP (mg/L) before and after treatment.
Changes in erythrocyte sedimentation rate (ESR). | Baseline, 4 weeks and 12 weeks
  Evaluating changes in concentration of ESR (mm/h) before and after treatment.
Changes in serum lipopolysaccharide-binding protein (LBP) | Baseline, 4 weeks and 12 weeks
  Evaluating changes in LBP concentration in serum before and after treatment.
Changes in serum intestinal fatty acid-binding protein (I-FABP) | Baseline, 4 weeks and 12 weeks
  Evaluating changes in I-FABP concentration in serum before and after treatment.
Changes in serum soluble cluster of differentiation 14 (sCD14) | Baseline, 4 weeks and 12 weeks
  Evaluating changes in sCD14 concentration in serum before and after treatment.
Numbers of participants with treatment-related adverse events | 12 weeks
  Adverse effects include fever, rash, abnormal liver and kidney function, new-onset infection, and any abnormal measures associated with experimental drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China